CLINICAL TRIAL: NCT05488015
Title: Effects of Global Postural Re-education (GPR) on Stress and Sleep Quality in Health Science Teachers and Students
Brief Title: Effects of GPR on Stress and Sleep Quality in Health Sciences
Acronym: GPRstress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/2021
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-08

CONDITIONS: Stress, Psychological
Keywords: Cortisol; Sleep quality; students; lecturers; self-treatment
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor responsible for collecting the results was blinded, without commenting on the group from which the patient came.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1 week of familiarisation through videos, audios and information documents, followed by 8 weeks of self-treatment with two GPR postures.
  Interventions: Other: Global Postural Re-education (GPR)
- Control (Active Comparator): No change in lifestyle habits during the 8-week trial.
  Interventions: Other: Lifestyle habits

INTERVENTIONS:
Other: Global Postural Re-education (GPR) — GPR intervention lasted 8 weeks. Each week the postures had to be performed on 4 or 5 days.
  Other Names: GPR
  Arms: Intervention
Other: Lifestyle habits — No change in lifestyle habits during the 8-week trial.
  Other Names: Normal life
  Arms: Control

SUMMARY:
Stress is a physiological reaction of our organism to situations that are perceived as threats. Of the different types of stress, emotional stress understood as a feeling of tension in difficult and unmanageable situations is increasingly prevalent in the western population and is responsible for a multitude of physical and psychological health disorders. In the same vein, sleep is a process experienced with a circadian (daily) periodicity in which there is a direct detachment from the environment and is necessary to maintain physiological, psychological and/or behavioral activities correctly.

Both teachers and students in higher education are examples of populations in which emotional stress and problems related to sleep quality have been described, with women being more sensitive to these problems.

The beneficial effects of physical exercise on different cognitive variables have been described, and it has been possible to characterise these effects on the physiological triggers of stress and sleep and, therefore, on alterations in the nervous and hormonal systems. Along these lines, Global Postural Re-education (GPR) is a physical therapy designed to re-establish the coordination of muscle chains and relieve pain. It has been established that GPR is a therapy in which the active participation of the patient is necessary so that it can be framed as physical exercise, with a structured execution protocol.

The overall aim of this study is to test whether a self-treatment therapy with RPG, after a learning and familiarisation phase, performed for 8 weeks, can have positive effects on stress reduction and improvement of sleep quality in female teachers and students of health sciences.

DETAILED DESCRIPTION:
The general objective of this study is to verify if a self-treatment therapy with GPR, after a learning and familiarization phase, carried out for 8 weeks, can have positive effects in reducing stress and improving sleep quality in teachers and health sciences students.

Intervention: GPR postures

1. Coxofemoral opening with closed arms or commonly called ground frog:

   The goal of this pose is to stretch the anterior muscle chain. The initial position of the patient is lying supine (face up) on the floor with the arms stretched out crosswise (abduction 90º) and the palms of the hands supinated (looking towards the ceiling). Feet together on the soles and knees apart. The lower back must remain in a neutral lordosis and pelvis at all times. The shoulders should be relaxed and away from the ears, that is, there should be no elevation of them, and the patient should have a sense of self-growth.
2. Hip closure with closed arms or commonly called frog in the air:

The objective of this posture is to make a global stretch of the posterior muscular chain. The patient's initial position is lying supine on the floor with hip and knee flexion, for which they had to support their feet on a wall. When lying on the floor, the patient must be as close to the wall as possible to be able to perform the posture correctly. The soles of the feet should contact each other and be closest to the gluteal area. The upper limbs must be in 90º abduction with supination of the hands. The lower back must remain in a neutral lordosis and pelvis at all times. The shoulders should be relaxed and away from the ears, that is, they should not rise, and the patient should have a sense of growth.

A very important point is the breathing used during the performance of the postures. Inspiration should be performed by inflating the abdominal area. On expiration, air should be exhaled through the mouth, without pursing the lips, feeling how the sternum sinks and then the ribs close. It is very important to do it this way throughout the stretch.

Stress

Cortisol

Cortisol is a lipid molecule that allows the body to maintain itself in a state homeostatic. In addition, it performs important functions in metabolic systems, cardiovascular and immunological Cortisol secretion varies throughout the day. In relation to circadian rhythms, cortisol levels are higher in the morning than in the afternoon. Therefore, the normal cortisol curve will reach maximums in the early hours of the day and minimums during the last hours. The body reacts to stress by releasing chemicals into the body, including glucocorticoids. Cortisol is the main glucocorticoid in the zona fasciculata of the human adrenal cortex, therefore, high levels of stress will produce a high level of cortisol secretion, thus modifying the normal cortisol curve. Cortisol flows through the acini of the salivary glands and its concentration does not varies depending on the salivary flow. It has been shown that the measurement of salivary cortisol corresponds to that of serum cortisol, therefore, the collection of cortisol in saliva It is a non-invasive and simple method to measure free cortisol.

"Salivette® Cortisol from the brand "Sarstedt", was chosen as the method for hygienic collection of saliva from the different participants, and subsequent measurement of cortisol levels as indicator of stress levels. Participants can easily and autonomously collect saliva samples from home. The collection process was explained to them in detail, both in person and in writing (leaflets). Salivette® Cortisol consists of a plastic tube, inside which there is another smaller tube, which contains a cotton swab of biocompatible synthetic fiber, which allows a great absorption capacity and subsequent recovery of saliva by means of centrifugation. For the collection of the sample, the participants had to meet certain standards, such as: the cotton inside the small tube cannot be touched, but must be inserted directly to the mouth. It cannot be bitten, it must be moved by making circles inside from the mouth for 1 minute. And finally, it must be returned to the small tube of the same way that it is extracted, without touching it with the hands. In addition, for the collection of the sample, you cannot eat, drink, or brush your teeth when least 30 minutes before. Four samples were collected at different times of the day in order to establish the circadian rhythm of cortisol. The hours at which saliva should be collected were: upon waking (where the maximum levels of cortisol in saliva are reached), at 11:00 am, at 15:00 pm (concentration is the most linear) and at bedtime ( where the levels are minimum). The samples collected from this method by the participants were initially kept in the freezer of their homes. The following days, they were asked to take them to the Francisco de Vitoria University, where they were collected thanks to the collaboration of the Department of Physiotherapy, and stored in the refrigerator at 4ºC, before being transferred to the freezer of the Biotechnology laboratory, where they were stored. They were kept at a temperature of -80 ºC, until the moment of their analysis. This was carried out with the "CORTISOL Saliva ELISA SA E-6000" kit of the LDN® brand (48), which is specifically developed and approved to quantitatively measure cortisol in saliva in humans.

State-Trait Anxiety Questionnaire (STAI)

This questionnaire was designed in 1973 by Spielberger et al. in California. Subsequently, in 1989, it was adapted into a Spanish version by Seisdedos. The questionnaire represents one of the most widely used diagnostic tests, one of the first validated and sensitive to assess anxiety in the international clinical community. Stress and anxiety are closely related. While stress is an adaptation to the environment, anxiety is one of the most frequent emotional reactions caused by stress. As a consequence of stress, the measurement of anxiety through the STAI questionnaire was included in the present study. Exactly, two facets of anxiety are valued. The first, trait anxiety (A-R), which refers to the personal factors that intervene in capturing the anxiety level of the stimuli that are perceived. That is, a person with a higher A-R will perceive a stimulus as more threatening than a person with lower levels of A-R, thus characterizing individuals with a tendency to conceive different situations as hostile. The second facet, state anxiety (A-E), in relation to environmental stimuli, which are capable of triggering an anxiety response in the subject.

To measure both states, the questionnaire consists of two independent scales of self-assessment, each of which contains 20 items. Each item has 4 response possibilities, with 0 being nothing, 1 somewhat, 2 quite a bit and 3 a lot (49).

The points obtained from both scales can vary between 0 and 60. It can be distinguished as follows: in the low anxiety group, scores less than 9 for the STAI-State (STAI-E) and 11 for the STAI-Trait (STAI-R), and on the other hand, in the high anxiety group, scores greater than 26 for the STAI-E and 30 for the STAI-R.

Sleep Quality

Actigraphy The first measurements on sleep were taken based on the electrical activity of the sleeping human brain, using polysomnography, in the laboratory. In polysomnography, an electroencephalogram is used to study brain activity, electromyography for muscle spasms, and even eye movements are studied. Over time, other types of mechanisms have been studied to be able to carry out a sleep study under normal conditions and outside the laboratory, such as actigraphy, which uses an external means by means of a bracelet placed on the hand that measures activity during sleep. 24 hours. Actigraphy is a good physiological measure of sleep.

The activity wristbands used to take physiological measurements of sleep quality were the actigraph GT3X (55). The participants were instructed to wear the bracelet during the week before and after the intervention. They were instructed that they had to wear a full week at each intake (first week of the study and last) and, following the protocols for use of the brand, they were instructed that they could only remove the bracelet in all activities that implied the possibility of let them get wet In addition, the bracelet had to be worn on the non-dominant hand. To obtain the data from the bracelets, a Windows computer with Actilife version 6.9 software (58) was used. The data thrown by the bracelets are In Bed (time to go to bed), Out Bed (time to get up), latency (time that passes from going to bed until falling asleep in minutes), Efficiency (the efficiency of sleep itself, according to the hours that slept and those in bed), Total Time in Bed, TST (Total Sleep Time - total sleep time expressed in minutes), WASO (Wake After Sleep Onset - wake-up time while sleeping), # of Awakenings (Number of awakenings in the night) and Avg Awakening (Average time of each awakening in the night).

Pittsburgh Sleep Quality Index

The Pittsburgh Sleep Quality Index (PSQ1) was designed by Bruysse et al in 1988, with the aim of having a measurement instrument for the quality of sleep, later this version was adapted. It is a self-administered questionnaire consisting of 19 self-assessed items and 5 evaluated by the bed partner.

These items provide information on 7 aspects related to sleep, such as:

* Subjective sleep quality.
* Sleep latency.
* Duration of sleep time.
* Usual sleep efficiency.
* Sleep disturbances.
* Use of sleep medications.
* Diurnal dysfunction. The first 4 questions are answered concretely, in the following ones it is possible to obtain a score from 0 to 3. Where 0 represents no difficulties and 3 severe difficulties.

To obtain the final score, only the first 18 questions are evaluated, which are the ones that must be answered by the subject himself (the last 5 should be answered by the bed partner) adding add each of the 7 items. It was considered that a score equal to or greater than 6 represents a poor quality of sleep.

Sleep Diary

The Sleep Diary was included as an instrument to complement the information collected through the PSQ1 questionnaire, previously explained, and to be able to evaluate and carry out a more exhaustive follow-up of the effects of the intervention on sleep quality. This was used as a self-monitoring tool that allowed us to subjectively estimate different parameters of interest in relation to sleep, such as: TST (total sleep time), SOL (nocturnal sleep onset latency), WASO (wake after onset ofsleep) and perceived sleep quality or satisfaction using the Likert scale established from 0 (very poor) to 4 (very good). The Central Consensus Dream Journal (CSD) consists of 9 items (which were translated into Spanish) that represent the most important parameters important:

1. Bedtime
2. Moment in which the subject tries to fall asleep.
3. Sleep onset latency.
4. Number of awakenings.
5. Duration of awakenings.
6. Final awakening time.
7. Time when you get up from bed.
8. Sleep quality.
9. Additional comments. It was delivered in Excel format to the participants, so that they could easily fill in every day as soon as possible after waking up, from the beginning to the end of the session.

intervention.

App "My Menstrual Calendar"

The menstrual cycle consists of a series of changes in the female genital tract, mainly in the ovary and uterus, being able to differentiate between the ovarian cycle and the uterine, endometrial or menstrual. These changes begin with puberty, are repeated cyclically with periods that range between 20 and 38 days, the usual duration being 28 days, and ending with the arrival of the climacteric. The following phases can be differentiated in the ovarian cycle:

1. Follicular or preovulatory phase (day 1-13): hormone peaks are observed in this phase follicle-stimulating hormone (FSH) and estrogen, which reaches its maximum value 48 hours before the ovulation.
2. Ovulation (day 13-15): period in which the release of the egg occurs. What As a result of this process, a new endocrine tissue is developed, called the corpus luteous or yellow.
3. Luteal or postovulatory phase (day 15-25): if the fertilization process does not take place, an increase in the release, by the corpus luteum, of progesterone is observed. Environment On day 25, there is a drop in the concentration of ovarian hormones, giving rise to menstruation.

As a control, due to the great variation within the cycle of the different hormones, decided to track the menstrual cycle of the participants during the months of intervention, allowing us to estimate in which phase of the cycle they were during the days Cortisol samples were taken, and the questionnaires used in the study were filled out.

study, PSQ1 and STAI. As can be seen in the study by Wilson M.C et al., there are you still doubt whether cortisol levels vary depending on the phase of the cycle in which is the woman, especially in the luteal phase, so it is of interest to have with this variable, as a backup to possible alterations when analyzing the data by part of the researchers. Similarly, it has been seen that the quality of sleep can also be affected depending on gender. Sleep disorders, anxiety and depression are more prevalent in women and represent a health problem. More women report complaints of insomnia, insufficient sleep, or poor subjective quality of sleep. These complaints are usually more frequent after puberty, or at different times such as pregnancy or menopause, so it could be due to hormonal events.

For all this, due to the relationship between anxiety, sleep quality and sexual hormones It is interesting as a control, to keep track of the menstrual cycle during the months of intervention. For this, the participants used the application called "My Menstrual Calendar". It is a free and easy-to-use application, where participants had to enter the exact days of their menstrual period during the two months of interest, as well as information on how they felt on those days.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-45 years
* Health sciences students and teachers.

Exclusion Criteria:

* Rotating work shifts
* Pregnant
* Use of medications (Non-steroidal anti-inflammatory drugs (NSAIDs)
* Acute or subacute back pain
* Musculoskeletal and neurological injuries associated with sleep disorders
* Sleep disorders (sleep apnea, circadian rhythm sleep disorder)
* Tumor, rheumatological, adrenal or pituitary diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Cortisol | Changes along the day from wake-up to time to bed during 8 weeks
  Cortisol concentrations are measured by saliva swab in the study patients.
State-Trait Anxiety Inventory Trait (STAI-T) | At the beginning of procedure and at the end (8 weeks)
  Anxiety is one of the most frequent emotional reactions caused by stress. Anxiety has been used to measure stress levels through the State and Trait Anxiety Questionnaire (STAI).The range of possible scores for the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
State-Trait Anxiety Inventory State (STAI-S) | At the beginning of procedure and at the end (8 weeks)
  Anxiety is one of the most frequent emotional reactions caused by stress. Anxiety has been used to measure stress levels through the State and Trait Anxiety Questionnaire (STAI). The range of possible scores for the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Pittsburgh Sleep Quality Index (PSQI) | At the beginning of procedure and at the end (8 weeks)
  The PSQ1 is a validated questionnaire consisting of 19 self-assessed items plus 5 items assessed by the bed partner or roommate. It provides information on 7 sleep-related aspects: subjective sleep quality, sleep latency, sleep time duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, daytime dysfunction. The first 4 questions are answered concretely, and the following questions can be scored on a 4-point scale (0-3).

SECONDARY OUTCOMES:
Wakefulness After the Onset of Sleep (WASO) | At the beginning of procedure and at the end (8 weeks)
  One of the variables of the sleep diary (actigraphy). WASO is defined as the minutes awake during the sleep period after sleep onset (the first 2 continuous minutes scored as sleep). Sleep efficiency, defined as the percent of time scored as sleep during the sleep period, was examined as a continuous variable and using the cutpoint <70%.
Sleep efficiency (SE) | At the beginning of procedure and at the end (8 weeks)
  One of the variables of the sleep diary (actigraphy). SE can calculate by dividing the time asleep by the total time in bed. So, if a subject sleep for six out of eight hours in bed, the sleep efficiency is 75%. Scores of 85% or higher is considered "normal." Scores below 60% is considered "sleep no effective".
Total Sleep Time (TST) | At the beginning of procedure and at the end (8 weeks)
  One of the variables of the sleep diary (actigraphy). The overall sleep score is a sum of the individual scores in sleep duration, sleep quality, and restoration, for a total score of up to 100. Most people get a score between 72 and 83. Sleep score ranges are: Excellent: 90-100.
Sleep Onset Latency (SOL) | At the beginning of procedure and at the end (8 weeks)
  One of the variables of the sleep diary (actigraphy). The basic approach of the MSLT is that lower scores indicate greater sleepiness and vice versa. It is accepted that a mean score of less than 5 min indicates a pathological level of daytime sleepiness. This level is associated with impaired performance in patients and in sleep-deprived normal subjects. Adult normal controls usually range from 10 to 20 min. Scores between 5 and 10 min indicate moderate sleepiness and may or may not be pathological.
Awakenings | At the beginning of procedure and at the end (8 weeks)
  This variable was measured by means of a bracelet that counts the number of times the subject wakes up during the night. A high number of awakenings indicates poor sleep quality, while no awakenings is the best rating of sleep quality.
Awakenings average | At the beginning of procedure and at the end (8 weeks)
  This variable was measured by means of a bracelet in which the number of times the subject wakes up during the night is counted and an average is taken to count the number of times a subject has woken up over a period of time in order to make an assessment of the quality of sleep. A high number of awakenings average indicates poor sleep quality, while value of 0 is the best rating of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: David Varillas Delgado, PhD, Study Director — Universidad Francisco de Vitoria, crta Pozuelo-Majadahonda km 1.800 PC 28223, Madrid, Spain
Locations (1):
- David Varillas Delgado, Pozuelo de Alarcón, Madrid, Spain

REFERENCES:
- [Derived] Rodriguez-Aragon M, Varillas-Delgado D, Gordo-Herrera J, Fernandez-Ezequiel A, Moreno-Heredero B, Valle N. Effects of global postural re-education on stress and sleep quality in health sciences female students: a randomized controlled trial pilot study. Front Psychiatry. 2024 Aug 28;15:1404544. doi: 10.3389/fpsyt.2024.1404544. eCollection 2024. PMID 39262580